CLINICAL TRIAL: NCT00329992
Title: Brief Eclectic Psychotherapy for PTSD - a Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Herrmann-Klaus-Stiftung, Switzerland (Unknown); Olga Mayenfisch Stiftung, Zurich, Switzerland (Unknown); Jubiläumsspende für die Universität Zürich, Switzerland (Unknown)
Responsible Party: Prof. Ulrich Schnyder, MD, University Hospital Zurich, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3200BO-102204
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): 16 sessions Brief Eclectic Psychotherapy
  Interventions: Behavioral: Brief Eclectic Psychotherapy for PTSD
- Control group (Placebo Comparator): Minimal attention waitlist group
  Interventions: Behavioral: Brief Eclectic Psychotherapy for PTSD

INTERVENTIONS:
Behavioral: Brief Eclectic Psychotherapy for PTSD — 16 weekly sessions (50min) of Brief Eclectic Psychotherapy for PTSD
  Other Names: BEP

SUMMARY:
Participants are randomly assigned to either 16 sessions of Brief Eclectic Psychotherapy (Gersons et al. (2000) Journal Trauma Stress 13: 333-348), comprising psychoeducation, exposure, mementos and writing assignments, domain of meaning and integration, farewell ritual, or a minimal attention control group that will be offered 16 sessions of BEP after a waiting time of four months. Participants in the minimal attention control group receive monthly telephone calls and complete a symptom self monitoring diary (Tarrier, N. et al. (1999) Behavior Therapy 30: 597-605) for three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clear memory of an "index" traumatic event (sufficient for constructing a scene to be used in exposure) that occurred no less than six months prior to entering the trial (Montgomery and Bech 2000)
* PTSD according to the DSM-IV, related to the index traumatic event, as measured with the CAPS: frequency ≥ 1 and intensity ≥ 2 for a symptom to be counted plus a minimum level of overall severity ≥ 50
* Not receiving other psychotherapy for PTSD during the 16 weeks of active treatment; psychotherapy for other problems, brief check-ins with an existing therapist, and attendance at self-help groups will be allowed
* If on psychoactive medication: on a stable medication regimen for a minimum of two months prior to entering the trial
* Aged between 18 and 70 years
* Sufficient proficiency in the German language to participate in BEP
* Consent to be randomized into the trial

Exclusion Criteria:

* Current psychotic, bipolar, substance-related, or severe personality disorder
* Current severe depressive disorder
* Severe cognitive impairment or a history of organic mental disorder
* Evidence of PTSD or depression immediately prior to the index trauma
* Ongoing threat of traumatic exposure
* Prominent current suicidal or homicidal ideation
* Asylum seeking status

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-04; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity (CAPS, Blake et al. 1998; Post-therapy / post-waitlist comparison, controlled for baseline scores | Last month

SECONDARY OUTCOMES:
Ability to work and use of health care facilities | Last months
Comorbidity: Structured Clinical Interview for DSM-IV SCID I (First et al. 1996); Hospital Anxiety and Depression Scale HADS (Zigmond and Snaith 1983) | Last month
Questions on Life Satisfaction FLZ (Henrich and Herschbach 2000) | Last month
Posttraumatic Cognitions Inventory PTCI (Foa et al. 1999) | Last month
Posttraumatic Growth Inventory PGI (Tedeschi and Calhoun 1996) | Since trauma
EEG, event-related potentials: P300 | At assessment
Post-therapy / post-waitlist comparison, follow-up at 6month post therapy | Last month

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schnyder, MD, Principal Investigator — University of Zurich; Lutz Wittmann, MA, Principal Investigator — University of Zurich
Locations (1):
- Psychiatric Department, University Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Schnyder U, Muller J, Maercker A, Wittmann L. Brief eclectic psychotherapy for PTSD: a randomized controlled trial. J Clin Psychiatry. 2011 Apr;72(4):564-6. doi: 10.4088/JCP.10l06247blu. No abstract available. PMID 21527127